CLINICAL TRIAL: NCT00417989
Title: The STAR 3 Study - A Prospective, Randomized, Two-Arm Study to Compare the Efficacy of the MiniMed Paradigm REAL-Time System Versus Multiple Daily Injections (MDI) in Subjects Naïve to Insulin Pump Therapy
Brief Title: Study to Compare Efficacy of the MiniMed Paradigm REAL-Time System Vs. MDI in Subjects Naive to Insulin Pump Therapy
Acronym: STAR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP179/Z25
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2011-03-10 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes
Keywords: Glycemic control; Sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 722 sensor augmented pump (Experimental): 722 arm: MiniMed Paradigm REAL-Time System using NovoLog/NovoRapid for 1 year
  Interventions: Device: MiniMed Paradigm REAL-Time System
- Multiple Daily Injections (MDI) (No Intervention): MDI arm: Continue with current MDI therapy using Lantus and NovoLog/NovoRapid for 1 year

INTERVENTIONS:
Device: MiniMed Paradigm REAL-Time System — Paradigm 722 insulin pump Paradigm REAL-Time Transmitter Sensor ComLink Paradigm Link glucose meter
  Other Names: Medtronic Paradigm REAL-Time System
  Arms: 722 sensor augmented pump

SUMMARY:
Primary Outcomes: Average decrease in A1c from baseline to end of Study Phase (52 weeks) for subjects in the "722 Group" is greater than that for subjects in the "Control (MDI) Group".

Secondary Outcomes: Incidence and frequency of severe hypoglycemia; Measure of glycemic variability, Area Under the Curve (AUC); Quality of Life; and Health Economic Outcomes (MRU)

DETAILED DESCRIPTION:
Glycemic control remains a significant challenge for adult, adolescent and pediatric Type 1 diabetics. The current first line standard of care continues to be MDI therapy utilizing a long acting analog insulin. Continuous Glucose Monitoring (CGMS) is currently used by clinicians to record continuous, retrospective glucose measurements, which aid in identification of glycemic excursion patterns. This data is then used to make future therapy change recommendations. The MiniMed Paradigm REAL-Time System transmits real-time glucose measurements to the insulin pump every 5 minutes, allowing users to view their current glucose values, as well as to review glycemic excursions and trends over a 24-hour period. Additionally, data can be downloaded from the monitor to a personal computer, using appropriate software, so that the patient and physician can see a complete picture of glucose trends over time. The System will also alert users of high and low glucose levels, and allow subjects and their clinicians to treat to a therapeutic target HbA1c under carefully monitored conditions.

Subjects wearing the MiniMed Paradigm REAL-Time System will be compared to subjects that continue on their current MDI therapy, that includes a long acting analog insulin, over a 12 month period to evaluate changes in glycemic control (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 to 70 years
* Has been treated by the Principal Investigator or referring physician within the same practice for at least six months prior to screening
* Is fluent in speaking, reading and understanding English
* Has Type 1 diabetes mellitus, diagnosed by c-peptide, insulin antibodies, or prior documented DKA, or by a clinical picture consistent with Type 1 diabetes and excluding type 2 diabetes i.e. - previous ketosis as evidenced by laboratory evidence of urine ketones or alteration in bicarbonate levels with corresponding increased glucose levels, diagnosed at least 6 months prior to study entry, or has a fasting C-peptide that meet criteria of 110% of lower limit of normal or 200% of lower limit of normal in the presence of renal insufficiency (creatinine clearance < 50ml/min) at screening
* Is insulin infusion pump naїve or has not used an insulin pump within the last three years
* Currently is treated with insulin administration by injection > (greater or equal to) three (3) times daily and therapy has included the use of a long acting analog insulin for at least the previous 3 months prior to screening
* Performs fingerstick blood glucose (BG) testing an average of four times per day in the 30 days prior to screening
* Within 6 months prior to study entry and at Screening Visit 1, subject has a documented A1c level =/> 7.4% and =/< 9.5%

Exclusion Criteria:

* Is pregnant or planning to become pregnant during the course of the study
* Has suffered two or more documented events of severe hypoglycemia without warning of impending low glucose levels, within the previous 12 months
* Currently using oral or injectable steroids or immunosuppressant medications
* Use of any other pharmaceutical agent, other than insulin to treat diabetes, within the three months prior to screening;
* Has a current history of alcohol or drug abuse
* Has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), or thromboembolic disease in the 3 months prior to screening
* Has uncontrolled hypertension (diastolic blood pressure >100 mmHg and/or sustained systolic level [3 successive readings] > 160). Subjects who are taking antihypertensive medication will not be excluded provided they are maintained at a stable dose for 3 months prior to screening
* Has serious or unstable medical or psychological conditions (e.g., eating disorders, clinical depression, anxiety disorder) which, in the opinion of the Investigator, would compromise the subject's safety or successful participation in the study
* Is undergoing renal dialysis, including hemodialysis and continuous ambulatory peritoneal dialysis (CAPD)
* Has evidence of any allergic dermatological condition (e.g., severe adhesive sensitivity)
* Has recurrent episodes of skin infections or history of staphylococcus infection carrier state
* Has potential for lack of compliance or any other issue that may preclude the subject from satisfactory participation in the study, based on Investigatory judgment

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MD, Principal Investigator — University of Maryland, Baltimore; William V Tamborlane, MD, Principal Investigator — Yale University; Scott W Lee, MD, Study Director — Medtronic Minimed
Locations (30):
- United States (26):
  - Scripps Institute, La Jolla, California
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Barbara Davis Center, University of Colorado, Boulder, Colorado
  - Yale University, New Haven, Connecticut
  - Diabetes Research Institute (DRI), Miami, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Mid-America Diabetes Associates, Wichita, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Joslin Clinic, Boston, Massachusetts
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota International Diabetes Center, Saint Louis Park, Minnesota
  - Children's Hospital of St. Paul, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center Diabetes Research Clinic, Durham, North Carolina
  - Diabetes and Obesity Center, East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Utah Diabetes Center, Salt Lake City, Utah
  - University of Wisconsin Health West, Madison, Wisconsin
- Canada (4):
  - Endocrine Research, Inc., Vancouver, British Columbia
  - Health Science Center Memorial Hospital of Newfoundland, St. John's, Newfoundland and Labrador
  - Kingston General Hospital, Kingston, Ontario
  - Toronto General Hospital - UHN, Toronto, Ontario

REFERENCES:
- [Derived] Perkins BA, Halpern EM, Orszag A, Weisman A, Houlden RL, Bergenstal RM, Joyce C. Sensor-augmented pump and multiple daily injection therapy in the United States and Canada: post-hoc analysis of a randomized controlled trial. Can J Diabetes. 2015 Feb;39(1):50-4. doi: 10.1016/j.jcjd.2014.03.003. Epub 2014 Aug 29. PMID 25175313
- [Derived] Bergenstal RM, Tamborlane WV, Ahmann A, Buse JB, Dailey G, Davis SN, Joyce C, Peoples T, Perkins BA, Welsh JB, Willi SM, Wood MA; STAR 3 Study Group. Effectiveness of sensor-augmented insulin-pump therapy in type 1 diabetes. N Engl J Med. 2010 Jul 22;363(4):311-20. doi: 10.1056/NEJMoa1002853. Epub 2010 Jun 29. PMID 20587585

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Daily Injection (MDI): MDI arm: Continue with MDI using Lantus and NovoLog/NovoRapid for 1 year
Period: Overall Study
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Started | 244 (Intent to Treat include safety population & subjects with baseline & 1 post baseline A1C measurement) | 241
Completed | 224 | 219
Not Completed | 20 | 22
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 0 | 1
Not completed — Physician Decision | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI) | Total
Number analyzed (Participants) | 244 | 241 | 485
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (17.47) | 31.50 (16.50) | 31.90 (16.98)
Age, Customized [Number; unit: participants]
  <=18 years | 77 | 72 | 149
  Between 19 and 70 years | 167 | 169 | 336
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 107 | 211
  Male | 140 | 134 | 274
Region of Enrollment [Number; unit: participants]
  United States | 216 | 211 | 427
  Canada | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c From Baseline to 52 Weeks
Description: Change is defined as A1c at Week 52 minus A1c at Baseline in each study arm. The difference between the change in each group will then be analyzed. A1c measure is defined as the percent of glycated hemoglobin using one standardized assay for all subjects.
Time Frame: Baseline and 52 weeks
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 244 | 241
Percent glycated hemoglobin | -0.8 (0.84) | -0.2 (0.89)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Null - There is no treatment group difference in A1c change from baseline to Week 52. Calculated that the enrollment of 495 patients would provide a power of 90% to detect an absolute difference of 0.35 percentage points in the primary outcome, assuming a SD of 1.2%; Test type: Non-Inferiority or Equivalence — Superiority test with margin of 0.35; p = 0.05, ANCOVA — Confidence Interval 95%; ANVOCA is adjusted by study group, gender, pooled site, continuous age, duration of diabetes, BMI, and Baseline glycated hemoglobin level (A1C); Mean Difference (Final Values) = 0.35, 95% CI 2-sided [0.24 to 0.46], Standard Deviation 1.2

2. Secondary Outcome: Difference in Frequency of Severe Hypoglycemia From Baseline to Week 52;
Description: Severe Hypoglycemia is defined as a hypoglycemic episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory Blood Glucose (BG) by finger stick of less than 50 mg/dL (2.8 mmol/L). The frequency evaluates the total number of events. This will be analyzed and compared between the two study arms from baseline to week 52.
Time Frame: Baseline and 52 weeks
Measure: Number; unit: number of events
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 244 | 241
number of events | 32 | 27

3. Secondary Outcome: Overall Difference in Rate of Severe Hypoglycemia Events Between Study Arms From Baseline to Week 52
Description: Severe Hypoglycemia is defined as a hypoglycemic episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory BG by finger stick of less than 50 mg/dL (2.8 mmol/L). The rate evaluates the number of participants that experienced at least one severe hypoglycemia event and compares this number between the two study arms from Baseline to week 52. This measure identifies the rate or frequency of unique participant events.
Time Frame: Baseline and 52 weeks
Measure: Number; unit: participants
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 244 | 241
participants | 21 | 17
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Superiority or Other; p = 0.84, Mantel Haenszel; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.64 to 2.41], Standard Deviation 2

4. Secondary Outcome: Changes in Hypoglycemia Area Under the Curve (AUC) From Baseline to Week 52;
Description: Hypoglycemia is defined as a recorded blood glucose event <70mg/dL. The amount of time spent below this parameter will be analyzed and compared between groups from Baseline to Week 52.
Time Frame: Baseline and 52 weeks
Measure: Mean (Standard Deviation); unit: mmol/dl*min
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 244 | 241
mmol/dl*min | 0.0 (0.66) | 0.0 (0.60)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Non-Inferiority or Equivalence — No power calculation based on this endpoint. Results will be calculated on testing for statistical difference between arms; p = 0.05, ANCOVA; ANVOCA is adjusted by study group, gender, pooled site, continuous age, duration of diabetes, BMI, and Baseline AUC

5. Secondary Outcome: Changes From Baseline in Hyperglycemia Area Under the Curve (AUC) From Baseline to Week 52
Description: Hyperglycemia is defined as a recorded blood glucose event > 180 mg/dL. The amount of time spent above this parameter will be analyzed and compared between groups from Baseline to Week 52.
Time Frame: Baseline and 52 weeks
Measure: Mean (Standard Deviation); unit: mmol/dl*min
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 244 | 241
mmol/dl*min | -11.9 (19.31) | -1.1 (22.07)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.05, ANCOVA; ANVOCA is adjusted by study group, gender, pooled site, continuous age, duration of diabetes, BMI, and Baseline AUC

6. Secondary Outcome: Quality of Life - Hypoglycemia Fear Scale (HFS), Overall Score
Description: Difference of Baseline and 52 Weeks in Hypoglycemia Fear Scale (HFS) Overall Score between the two study arms (adult subjects only) is presented. Both baseline and 52 weeks scores range from 0-100, with lower scores suggest higher satisfaction. Therefore, a negative number in the difference suggests higher satisfaction at 52 Weeks than Baseline.
Time Frame: Baseline and 52 weeks
Population: Adult population (18 and older) only
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 152 | 151
participants | -9.0 (16.04) | -2.4 (15.88)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -6.5, 95% CI [-9.760 to -3.273], Standard Deviation 16.0

7. Secondary Outcome: Health Economic Outcome
Description: Health Economic Outcome was a cost-effectiveness analysis combining estimates from the trial and the literature to populate the previously validated Center for Outcomes Research (CORE) Diabetes Model. Results represent the use of 3-day sensors. This analysis was restricted to only adult subjects (Age 19 to 70), therefore the number of participant analyzed is different. The goal was to estimate the long term cost effectiveness of Sensor Augmented Pump therapy from the perspective of the US health care system. The unit of measurement was cost in $ per year for sensor augmented pump group and MDI group. No formal statistical analysis was planned or performed
Time Frame: Baseline and 52 weeks
Measure: Number; unit: $
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 166 | 163
$ | 10,760 | 5,072

8. Secondary Outcome: Quality of Life - Short Form-36 (SF-36v2™), General Health
Description: Difference of Baseline and 52 Weeks in Short Form-36 (SF-36v2™), General Health, between the two study arms (adult subjects only) is presented. Both baseline and 52 weeks scores range from 0-100, with higher scores suggest higher satisfaction. Therefore, a positive number in the difference suggests higher satisfaction at 52 Weeks than Baseline.
Time Frame: Baseline and 52 Weeks
Population: Adult population (18 and older) only
Measure: Mean (Standard Deviation); unit: Participants
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 153 | 151
Participants | 2.7 (8.07) | -0.3 (7.13)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Superiority or Other; Mean difference; Mean Difference (Final Values) = 3.0, Standard Deviation 7.75

9. Secondary Outcome: Quality of Life - Insulin Delivery System Rating Questionnaire (IDSRQ) for Subject Satisfaction With Type of Insulin Therapy
Description: Difference of Baseline and 52 Weeks in Insulin Delivery System Rating Questionnaire (IDSRQ) for Subject Satisfaction with Type of Insulin Therapy, between the two study arms is presented. Both baseline and 52 weeks scores range from 0-100, with higher scores suggest higher satisfaction. Therefore, a positive number in the difference suggests higher satisfaction at 52 Weeks than Baseline.
Time Frame: Baseline and 52 Weeks
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
Number analyzed (Participants) | 220 | 214
participants | 18.4 (25.61) | -0.2 (21.77)
Statistical Analysis 1: Comparison: 722 Sensor Augmented Pump vs Multiple Daily Injection (MDI); Test type: Superiority or Other; Mean Difference; Mean Difference (Final Values) = 18.6, Standard Deviation 25.53

ADVERSE EVENTS:
Arm/Group | 722 Sensor Augmented Pump | Multiple Daily Injection (MDI)
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/241
Serious Adverse Events (participants affected / at risk) | 32/244 | 30/241
Other Adverse Events (participants affected / at risk) | 96/244 | 49/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 722 Sensor Augmented Pump (N=244) | Multiple Daily Injection (MDI) (N=241)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 4 (4) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoglycemia (Severe Hypoglycemia) (Metabolism and nutrition disorders) | 15 (20) | 13 (15)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Severe Hypoglycemia) (Metabolism and nutrition disorders) | 8 (10) | 8 (12)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Diabetic Ketoacidosis (Ketoacidosis) (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Fibula Fracture (Fracture of Left Lower Leg, Fibula at Ankle) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Acute Gastroenteritis) (Infections and infestations) | 2 (2) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Non-Cardiac (Atypical) Chest Pain (General disorders) | 1 (1) | 0 (0)
Skin Laceration (Traumatic Laceration to Dorsum of the Right Foot with extensor Hallucis Longus Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast Cancer (Left Breast Cancer: Invasive Ductal Adenocarcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral Injury (Urethral Tear) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cellulitis (Cellulitis of Left Lower Leg) (Infections and infestations) | 2 (2) | 1 (1)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Limb Crushing Injury (Crush Injury to Right Lateral Thigh) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope Vasovagal (Syncope Vasovagal Response) (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Kidney Stones) (Renal and urinary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Did not meet protocol criteria for DKA
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Did not meet protocol definition of Severe Hypoglycemia
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 722 Sensor Augmented Pump (N=244) | Multiple Daily Injection (MDI) (N=241)
Hypoglycemia (Metabolism and nutrition disorders) | 32 (88) | 28 (56)
Infusion/application site infection/abscess (Infections and infestations) | 12 (13) | 1 (1)
Application site bleeding/bruising/irritation/pain (General disorders) | 20 (20) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 36 (51) | 17 (22)
Hyperglycemia (Metabolism and nutrition disorders) | 37 (46) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days